CLINICAL TRIAL: NCT03182699
Title: Effect of Etelcalcetide on Cardiac Hypertrophy in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effect of Etelcalcetide on Cardiac Hypertrophy in Hemodialysis Patients
Acronym: EtECAR-HD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rainer Oberbauer (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Rainer Oberbauer, Univ.-Prof. Rainer Oberbauer, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Etecarhd
Record Dates: First submitted 2017-05-31; First posted 2017-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease Requiring Chronic Dialysis; Left Ventricular Hypertrophy
Keywords: Secondary Hyperparathyroidism; Hemodialysis; Left Ventricular Hypertrophy; FGF 23; Etelcalcetide; Alfacalcidol
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypertrophy, Left Ventricular | interventions — Echocardiography; Clinical Laboratory Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Radiologist investigating the cMRI and physician performing the echocardiography will be blinded.
  Patients will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etelcalcetide (Experimental): Patients will receive Etelcalcetide i.v. 3 times per week after dialysis Dose titration will take plac every 4 weeks in the first 16 weeks Dose adaptation is based on PTH, SerumCa++, SerumPhosphate, T-50-time
  Interventions: Diagnostic Test: cardiac MRI; Diagnostic Test: echocardiography with strain; Diagnostic Test: Laboratory tests; Diagnostic Test: Body composition monitoring; Diagnostic Test: lung ultrasound
- Alfacalcidol (Active Comparator): Patients will receive Alfacalcidol i.v. 3 times per week after dialysis Dose titration will take plac every 4 weeks in the first 16 weeks Dose adaptation is based on PTH, SerumCa++, SerumPhosphate, T-50-time
  Interventions: Diagnostic Test: cardiac MRI; Diagnostic Test: echocardiography with strain; Diagnostic Test: Laboratory tests; Diagnostic Test: Body composition monitoring; Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: cardiac MRI — non contrast heart MRI at baseline and after 1 year of therapy
Diagnostic Test: echocardiography with strain — echocardiography at baseline and after 1 year of therapy
Diagnostic Test: Laboratory tests — drawing blood from dialysis machine
Diagnostic Test: Body composition monitoring — Measurement with BCM (Fresenius) machine
Diagnostic Test: lung ultrasound — ultrasound

SUMMARY:
Background:

Calcimimetic therapy has been shown to reduce systemic FGF23 levels, which themselves are associated with left ventricular hypertrophy (LVH) in chronic kidney disease (CKD).

Methods/design:

This is a randomized multicenter trial in which the effect of etelcalcetide in comparison to alfacalcidol on LVH and cardiac fibrosis in hemodialysis patients with secondary hyperparathyroidism (sHPT) will be investigated.

The investigators will perform a comparative trial testing etelcalcetide vs. alfacalcidol treatment on top of conventional HPT therapy for 12 months. A total of 62 hemodialysis patients with sHPT and LVH will be enrolled in the study. After a washout of all calcimimetic and vitamin D treatment, subjects will be randomized at 1:1 ratio to either etelcalcetide or alfacalcidol. The participants will undergo cardiac imaging consisting of cardiac resonance imaging (cMRI) and strain echocardiography before and at baseline and one year. Etelcalcetide or alfacalcidol will be administered intravenously three times per week following chronic hemodialysis treatment.

The primary end point will be a change in left ventricular mass index (LVMI) measured in g/m2. As secondary end points the changes in left atrial diameter (LAD), cardiac fibrosis, wall motion abnormalities and left ventricular function, changes in serum FGF 23 and soluble Klotho levels as well as changes in proBNP as well as pre- and postdialysis troponin T (TnT) levels will be determined. Additionally a quantitative analysis of the treatment influence on the individual metabolites of the renin-angiotensin-aldosterone system (RAAS) will be performed using mass spectrometry ("RAAS fingerprint").

DETAILED DESCRIPTION:
Hypothesis and specific aims

In this randomized multicenter trial the investigators will study the effect of etelcalcetide in comparison to alfacalcidol on left ventricular hypertrophy and fibrosis in hemodialysis patients with secondary hyperparathyroidism (sHPT). Etelcalcetide is a calcimimetic drug that has been approved for the treatment of secondary HPT in hemodialysis patients.

Fibroblast growth factor 23 (FGF23) levels rise early in the development of chronic kidney disease (CKD) and recent studies have shown that FGF23 increases the development of left ventricular hypertrophy in these patients. Elevated FGF 23 levels are further associated with progression to end-stage renal disease, cardiac events and all-cause mortality. In animal models a blockade of FGF23 ameliorates the pathologic effect on left ventricular mass and function. Calcimimetic therapy has been shown to reduce systemic FGF23 levels, while vitamin D therapy is known to elevate FGF23. However, there is limited data on the clinical relevance of therapeutic modification of FGF23 levels in humans.

The investigators specifically hypothesize that treatment with etelcalcetide ameliorates pathological changes in cardiac structure in dialysis patients with sHPT by suppression of systemic FGF23 levels.

Specific aim 1

In this trial the investigators will determine the influence of calcimimetic therapy on left ventricular hypertrophy (LVH) in hemodialysis patients with sHPT: They will perform a head-2-head trial testing etelcalcetide vs. alfacalcidol treatment on top of conventional HPT therapy (phosphate binders, calcium supplementation and if necessary vitamin D substitution or cinacalcet) for 12 months. Etelcalcetide or alfacalcidol will be administered intravenously three times per week following chronic hemodialysis treatment. The primary end point will be a change in left ventricular mass index (LVMI) that will be assessed using cardiac magnetic resonance imaging (cMRI) at baseline and after 12 months of treatment. As secondary end points we will measure changes in left atrial diameter (LAD), cardiac fibrosis (using T1 mapping and cardiac strain), wall motion abnormalities and left ventricular function (measured in cMRI and echocardiography), changes in serum FGF 23 and soluble Klotho levels as well as changes in proBNP as well as pre- and postdialysis troponin T (TnT) levels.

Specific aim 2

The pathophysiology by which elevated FGF 23 levels can cause cardiac remodeling is still unresolved. The two major hypothesis propose either a direct effect of FGF 23 on the myocardium or a predominantly volume dependent effect caused by FGF 23 and Klotho mediated renal sodium retention:

* Sodium and volume balance in dialysis patients without residual renal function is regulated by ultrafiltration and not by renal sodium handling. In this trial the investigators will perform a stratified randomization procedure to ensure an equal distribution of dialysis patients with residual renal function and those without in both treatment groups.
* Additionally, FGF 23 directly inhibits Angiotensin converting enzyme 2 (ACE 2) as the central enzyme of the antifibrotic alternative renin-angiotensin-aldosterone system (RAAS) and shifting the RAAS toward the pro fibrotic Angiotensin II. To assess suppression of ACE 2 we will measure Ang 1-5 and Ang 1-7 levels by quantitative analysis of the individual metabolites of the RAAS using mass spectrometry ("RAAS fingerprint").

The specific design of this trial will therefore contribute to the fundamental understanding of FGF 23 mediated myocardial remodeling.

After completion of the trial two T-50-test will be performed in each patient from existing frozen serum samples (one at baseline and one at the end of 12 months of treatment). The measurement of the T50-time can evaluate an individual's risk for the development of vascular calcification

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Treatment with maintenance hemodialysis 3 times a week for ≥ 3 months and ≤3 years
* sHPT defined by

  * PTH levels obtained from the central laboratory of ≥300 pg/mL and no prior treatment with a calcimimetic drug, or
  * PTH levels obtained from the central laboratory of ≥300 pg/mL in patients under vitamin D treatment following a washout phase of 4 weeks
  * patients under treatment with cinacalcet who will be eligible following a washout phase of 4 weeks
* serum calcium (corrected for serum albumin) levels obtained from the central laboratory of ≥ 2.08 mmol/L
* Signs of LVH (increased myocardial thickness in the left ventricle, increased interventricular septum thickness i.e. ≥12mm) irrespective of signs of cardiac fibrosis in cardiac imaging (Echocardiography)
* State of optimal fluid composition i.e. reaching the individual dry weight as measured with the help of a Body Composition Monitor (BCM) (more see below under section 4.9.2). Pulmonary edema will be excluded with the help of lung ultrasound (lung comet tails).
* No substantial dose change of calcium supplements, phosphate binders, dialysate calcium, or active vitamin D for 4 weeks before screening

Exclusion Criteria:

* Unstable medical condition based on medical history, physical examination, and routine laboratory tests, or judged unstable in the investigator's opinion
* Significantly impaired left ventricular systolic function or significant, hemodynamically effective heart valve defects
* History of any illness, which in the investigator's opinion, might confound the results of the study or pose additional risk
* Anticipated parathyreoidectomy within 12 months after randomization
* Scheduled date for kidney transplant from a living donor
* Uncontrolled hyperphosphatemia
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Subject has known sensitivity or intolerance to any of the products to be administered for the purpose of this study
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures
* Subject is pregnant, or is of child-bearing potential and not using adequate contraceptive precautions although this is highly unlikely in patients on maintenance hemodialysis.
* Contraindications for MRI (implanted MR-Unsafe - objects that are significantly ferromagnetic and pose a clear and direct threat to persons and equipment within the magnet room)
* Overhydration as measured in BCM or visualized in lung ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass index | one year
  Change of LVMI from baseline after a year-long treatment with either etelcalcetide or alfacalcidol.
  Measurement of LVMI (g/m2) with the help of cMRI

SECONDARY OUTCOMES:
Cardiac structure | one year
  Difference in left atrial diameter measured by cMRI (mm)
Cardiac structure | one year
  Change in LVMI progression in either treatment group (%) measured in cMRI
Cardiac structure | one year
  Change in LAD progression in either treatment group (%) measured in cMRI
Cardiac structure | one year
  Difference in cardiac fibrosis (%) measured by cMRI and cardiac strain
Cardiac structure | one year
  Difference in the progression of cardiac fibrosis (%) measured by cMRI and cardiac strain
Cardiac structure | one year
  Differences in cardiac function (ejection fraction - %) measured in cMRI
Cardiac structure | one year
  Differences in wall motion abnormalities measured in cMRI (%)
Laboratory parameters | one year
  Changes in metabolites of the RAAS (pg/ml) using mass spectrometry ("RAAS fingerprint") under either treatment
Laboratory parameters | one year
  Change from baseline serum levels of FGF23 (RU/mL) under either drug
Laboratory parameters | one year
  Change from baseline serum levels of s-klotho (pg/mL) under either drug
Laboratory parameters | one year
  Change from baseline in PTH (ng/l) under either treatment
Laboratory parameters | one year
  Change from baseline in 25-OH-Vit-D (nmol/L) under either treatment
Laboratory parameters | one year
  Change from baseline in 1,25-(OH)2-Vit-D (pg/mL) under either treatment
Laboratory parameters | one year
  Change from baseline in serum phosphate (mmol/l) under either treatment
Laboratory parameters | one year
  Change from baseline in serum calcium (mmol/l) corrected for serum albumin under either treatment
Laboratory parameters | one year
  Changes from baseline in proBNP (pg/ml) in either medication group
Laboratory parameters | one year
  Changes from baseline in pre- and postdialysis TnT (ng/ml) in either medication group
T-50-time measurement | one year
  After completion of the trial two T-50-test will be performed in each patient from existing frozen serum samples (one at baseline and one at the end of 12 months of treatment). The measurement of the T50-time can evaluate an individual's risk for the development of vascular calcification
Laboratory parameters | One year
  Longitudinal change in serum levels of FGF23 in pg/mL from baseline.
Laboratory parameters | One year
  Longitudinal change in serum levels of PTH in ng/L from baseline.
Laboratory parameters | One year
  Longitudinal change in serum levels of calcium corrected for albumin in mg/dL from baseline.
Laboratory parameters | One year
  Longitudinal change in serum levels of s-klotho in pg/mL from baseline.
Laboratory parameters | One year
  Longitudinal change in serum levels of phosphate in mg/dL from baseline.
Laboratory parameters | One year
  Longitudinal change in serum levels of 25-OH-Vitamin-D in nmol/L from baseline
Laboratory parameters | One year
  Longitudinal change in serum levels of 1,25-(OH)2-Vitamin-D in pg/mL from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Oberbauer, Univ.Prof., Principal Investigator — Head of the department of Nephrology of the MUVienna; Matthias Lorenz, Priv.Doz., Principal Investigator — Head of the Dialysis center (WDZ)
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - Wiener Dialysezentrum, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dorr K, Kammerlander A, Lauriero F, Lorenz M, Marculescu R, Beitzke D. Effect of etelcalcetide versus alfacalcidol on left ventricular function and feature-tracking cardiac magnetic resonance imaging in hemodialysis-a post-hoc analysis of a randomized, controlled trial. J Cardiovasc Magn Reson. 2023 Nov 6;25(1):62. doi: 10.1186/s12968-023-00975-4. PMID 37932788
- [Derived] Dorr K, Reindl-Schwaighofer R, Lorenz M, Marculescu R, Beitzke D, Hodlmoser S. Etelcalcetide Inhibits the Progression of Left Atrial Volume Index Compared to Alfacalcidol in Hemodialysis Patients. Cardiorenal Med. 2023;13(1):332-341. doi: 10.1159/000533899. Epub 2023 Sep 20. PMID 37729887
- [Derived] Dorr K, Hodlmoser S, Kammer M, Reindl-Schwaighofer R, Lorenz M, Reiskopf B, Jagoditsch R, Marculescu R, Oberbauer R. Bone Specific Alkaline Phosphatase and Serum Calcification Propensity Are Not Influenced by Etelcalcetide vs. Alfacalcidol Treatment, and Only Bone Specific Alkaline Phosphatase Is Correlated With Fibroblast Growth Factor 23: Sub-Analysis Results of the ETACAR-HD Study. Front Med (Lausanne). 2022 Jul 6;9:948177. doi: 10.3389/fmed.2022.948177. eCollection 2022. PMID 35872799
- [Derived] Dorr K, Kammer M, Reindl-Schwaighofer R, Lorenz M, Marculescu R, Poglitsch M, Beitzke D, Oberbauer R. The Effect of FGF23 on Cardiac Hypertrophy Is Not Mediated by Systemic Renin-Angiotensin- Aldosterone System in Hemodialysis. Front Med (Lausanne). 2022 Apr 26;9:878730. doi: 10.3389/fmed.2022.878730. eCollection 2022. PMID 35559350
- [Derived] Dorr K, Kammer M, Reindl-Schwaighofer R, Lorenz M, Prikoszovich T, Marculescu R, Beitzke D, Wielandner A, Erben RG, Oberbauer R. Randomized Trial of Etelcalcetide for Cardiac Hypertrophy in Hemodialysis. Circ Res. 2021 May 28;128(11):1616-1625. doi: 10.1161/CIRCRESAHA.120.318556. Epub 2021 Apr 7. PMID 33825489
- [Derived] Dorr K, Kammer M, Reindl-Schwaighofer R, Lorenz M, Loewe C, Marculescu R, Erben R, Oberbauer R. Effect of etelcalcetide on cardiac hypertrophy in hemodialysis patients: a randomized controlled trial (ETECAR-HD). Trials. 2019 Oct 24;20(1):601. doi: 10.1186/s13063-019-3707-7. PMID 31651370